CLINICAL TRIAL: NCT03387501
Title: Efficacy and Safety of the Concentrate of Autologous Rich Plasma in Growth Factors in the Treatment of the Thin Endometrium in Patients Undergoing Transfer of Cryo-preserved Embryos: Clinical Trial II.
Brief Title: Concentrate of Autologous Rich Plasma in Growth Factors in the Treatment of the Thin Endometrium
Acronym: APTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sara Rafael Fernandez (Other)
Responsible Party: Sponsor-Investigator, Sara Rafael Fernandez, Head of Assisted Reproduction Laboratory, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APTE
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Infertility; Infertility, Female
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRGF (Experimental): Plasma rich in growth factors (PRGF) administration
  Interventions: Drug: Plasma rich in growth factors (PRGF-Endoret)

INTERVENTIONS:
Drug: Plasma rich in growth factors (PRGF-Endoret) — Intrauterine administration of PRGF

SUMMARY:
This study evaluate the percentage of women with thin endometrium who achieve an endometrial thickness equal to or greater than 7 mm after administration of PRGF (plasma rich in growth factors)

ELIGIBILITY:
Inclusion Criteria:

* Women who signed informed consent.
* Women who understand the Spanish language.
* Women under 42 years

Exclusion Criteria:

* Thrombopenia.
* Congenital or acquired uterine malformations that reduce embryo implantation or term gestation.
* Ovarian tumors.
* Benign uterine tumors require surgical treatment
* Local acute inflammatory diseases
* Patients with malignant tumors requiring chemotherapy.
* Patients with acute or chronic infectious or inflammatory diseases requiring active treatment with drugs that may interfere with implantation and gestation.
* Chronic treatment with NSAIDs (Nonsteroidal anti-inflammatory drugs)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Percentage of women who achieve an endometrial thickness equal to or greater than 7 mm | 3 days after administration of PRGF
  Measurement of the endometrial thickness by ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Rafael, PhD, Study Chair — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No